CLINICAL TRIAL: NCT01132183
Title: An Open Label, Balanced, Randomized, Two-treatment, Single-dose, Crossover, Bioequivalence Study of Divalproex Sodium Coated Particles in Capsules, 125 mg With Depakote® Sprinkle 125 mg in Healthy Human Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Divalproex Sodium Capsules(Sprinkle),125 mg of Dr. Reddy's Under Fasting Condition (Apple Sauce)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Mr. Indu Bhushan / Sr. Director R & D, Dr.Reddy's Laboratories Limited,
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-638/06
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Healthy
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Divalproex Sodium (Experimental): Divalproex Sodium Coated Particles in Capsules, 125 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Divalproex Sodium
- Depakote Sprinkle (Active Comparator): Depakote Sprinkle 125 mg capsules of Abbott Laboratories, USA
  Interventions: Drug: Divalproex Sodium

INTERVENTIONS:
Drug: Divalproex Sodium — Divalproex Sodium Coated Particles in Capsules, 125 mg of Dr. Reddy's Laboratories Limited
  Other Names: Depakote Sprinkle

SUMMARY:
An open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose, crossover, bioequivalence study of Divalproex Sodium coated particles in capsules 125 mg with Depakote® Sprinkle125 mg capsules in healthy, adult, human subjects under fasting conditions.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose, crossover, bioequivalence study of Divalproex Sodium Capsules (Sprinkle), 125 mg of Dr.Reddy's Laboratories Limited,comparing with that of Depakote® Sprinkle 125 mg capsules of Abbott Laboratories, USA in healthy, adult, human subjects under fasting conditions with an adequate washout period of 10 days.

The subjects were given a single oral dose of medication (test study or reference medication) . The capsule was opened and all the contents were sprinkled over a spoonful of applesauce without a spillage and administered to the subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria to be considered for inclusion into this study:

1. Subjects who will provide written informed consent.
2. Subjects must be healthy, adult, human beings within 18-45 years of age (both inclusive) weighing at least 50 kg.
3. Having a Body Mass Index (BMI) between 18.5 and 24.9 (both inclusive), calculated as weight in Kg/height in m2
4. Subjects must be of normal health as determined by medical history and physical examination performed within 21 days prior to the commencement of the study.
5. Subjects whose screening laboratory values are within normal limits or considered by the physician/investigator to be of no clinical significance.
6. Availability of the subject for the entire study period and willingness to adhere to the protocol requirements as evidenced by written informed consent.

Exclusion Criteria:

The subjects will be excluded based on the following criteria during screening and during the study

1. Subjects incapable of understanding the informed consent.
2. Subjects who have:

   1. Systolic blood pressure less than 90 mm of Hg or more than 140 mm of Hg
   2. Diastolic blood pressure less than 60 mm of Hg or more than 94 mm of Hg. Minor deviations (2-4 mm of Hg) at check-in may be acceptable at the discretion of the physician/investigator.
   3. Pulse rate below 50/min or above 100/min.
3. History of hypersensitivity or idiosyncratic reaction to Investigational drug products or any other related drugs.
4. Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function.
5. Consumption of grapefruit for the past ten days prior to the dosing day until the completion of the study.
6. Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking from 48 hours before dosing and during sampling period.
7. Subjects who have taken over the counter or prescribed medications and enzyme modifying or any systemic medication for during the last 7 and 30 days respectively before dosing.
8. Subj eets who have participated in any other clinical investigation using experimental drug/donated blood in past 90 days before the date of start of study.
9. Subjects with clinically significant abnormalities (such as Laboratory Findings,ECG, X-Ray, Drugs of abuse, Alcohol etc.,) and/or with significant diseases (such as HIV, HCV, Syphilis, Hepatitis B etc.,).
10. Female subjects who are pregnant or who are able (women with child bearing potential) to become pregnant during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2007-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: S Sai Krishna, MBBS, Principal Investigator — Bioserve Clinical Research Pvt. Ltd.
Locations (1):
- Bioserve Clinical Research Pvt. Ltd., Hyd, Andhra Pradesh, India